CLINICAL TRIAL: NCT03767400
Title: Dynamic Optical Coherence Tomography (D-OCT) Aging Study: A Preliminary Evaluation of Structural Differences Between Young and Aged Skin, Cellulite and Atrophic Acne Scars in Female Caucasian Subjects With Fitzpatrick Skin Types I-III Utilizing Non-invasive in Vivo D-OCT.
Brief Title: Dynamic Optical Coherence Tomography(D-OCT) Aging Study: A Preliminary Evaluation of Structural Differences Between Young and Aged Skin, Cellulite and Atrophic Acne Scars in Female Caucasian Subjects With Fitzpatrick Skin Types I-III Utilizing Non-invasive in Vivo D-OCT.
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: SCRIC18-OCT-01
Record Dates: First submitted 2018-12-05; First posted 2018-12-06 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Skin Care

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A - Young skin (18 - 30 years old): Assessments will be made after facial cleansing on areas being imaged utilizing VivoSight Dynamic Optical Coherence Tomography (D-OCT). Post-study D-OCT images will be processed with VivoSight software. Assessments of participant's overall photodamage and participant's appearance of fine lines/wrinkles will be measured.
  Interventions: Device: Skin Imaging; Other: Facial Cleanser
- Group B - Aged skin (55 - 75 years old): Assessments will be made after facial cleansing on areas being imaged utilizing VivoSight Dynamic Optical Coherence Tomography (D-OCT). Post-study D-OCT images will be processed with VivoSight software. Assessments of participant's overall photodamage and participant's appearance of fine lines/wrinkles will be measured.
  Interventions: Device: Skin Imaging; Other: Facial Cleanser
- Group C - Atrophic acne scars (18 - 75 years old): Assessments will be made after facial cleansing on areas being imaged utilizing VivoSight Dynamic Optical Coherence Tomography (D-OCT). Post-study D-OCT images will be processed with VivoSight software. Assessments of participant's overall photodamage and participant's appearance of fine lines/wrinkles will be measured.
  Interventions: Device: Skin Imaging; Other: Facial Cleanser

INTERVENTIONS:
Device: Skin Imaging — Non-invasive in vivo skin imaging will be taken with the VivoSight D-OCT and the measurements will be acquired post-study utilizing VivoSight software.
Other: Facial Cleanser — Participants will be instructed to remove all makeup from the face and cleanse the face with SkinMedica Facial Cleanser at least 15 minutes prior to investigator assessments and photography, and at least 30 minutes prior to use of D-OCT. Particiapnts in the cellulite group will have the thigh area cleansed with Facial Cleanser at least 15 minutes prior to photography and at least 30 minutes prior to use of D-OCT. For standardization, this procedure will be performed with SkinMedica Facial Cleanser (to remove makeup and cleanse the face and thigh (if applicable)) for all the participants.
  Other Names: SkinMedica® Facial Cleanser

SUMMARY:
This single-center clinical study is being conducted over the course of 2 weeks to conduct an exploratory pilot study as a preliminary evaluation of D-OCT's ability to measure skin changes from aging. Assess structural differences between young and aged skin on the face. To identify the structural characteristics of atrophic acne scars relative to normal skin on the face. To explore characteristics of cellulite relative to normal skin on the thigh in young and aged skin.

ELIGIBILITY:
Inclusion Criteria:

* Female Caucasian subjects with Fitzpatrick skin types I-III that meet one of the criteria listed below:

  1. Ages 18-30 years old without acne scars on the face with or without visible cellulite on posterior thigh, or
  2. Ages 55-75 years old without acne scars on the face with or without visible cellulite on posterior thigh, or
  3. Ages 18-75 years old with atrophic acne scars
* Subject has completed an appropriately administered informed consent process which includes signing the IRB approved consent form.
* Good general health and free of any disease state or physical condition (e.g. psoriasis, rosacea, scars, tattoos etc.) which, in the investigator's opinion, might impair evaluations of the test sites or expose the subject to an unacceptable risk by study participation.
* Willingness to remove all makeup on the day of the visit. Makeup may be applied after the study visit has been completed.
* Willingness to cleanse their face and remove all face makeup at each scheduled clinic visit. No other topical products should be applied to the face until the study visit has been completed.

  i. For cellulite subgroup, willingness to have thigh cleansed at each scheduled clinic visit.
* Willingness to have investigator exams, skin instrumentation measurements, and digital photos performed on the face and/or thigh (for cellulite subgroup).
* Women of childbearing potential must not be pregnant at the time of the study.

Exclusion Criteria:

* Has any condition that, in the opinion of the investigator, would make it unsafe for the subject to participate in the study or interfere with their clinical assessments (including conditions that require the concurrent use of anticoagulants, bleeding coagulopathies, photosensitivity diseases).
* Individuals with active symptoms of allergy, cold sore or warts, active psoriasis or eczema, rosacea, sunburn, open wounds, neurotic excoriations, tattoos, or other skin conditions in the test areas that would interfere with the assessments of this study.
* Individuals who are pregnant.
* Uncontrolled disease such as diabetes, hypertension, hyper or hypo-thyroidism, active hepatitis, immune deficiency, or autoimmune.
* Individuals who have a pre-existing or dormant dermatologic condition (e.g. history of severe psoriasis, atopic dermatitis, rosacea, skin cancer, etc.)
* Individuals who have routinely used any of the following topical products, prescription products, or had any of the listed treatments/procedures within the listed time frame prior to study entry or will use during study:

  1. Any product that the investigator deems that could affect the study objectives. These include products that address skin imperfections. This does not include a basic cleanser, moisturizer and sunscreen.(time frame 2 weeks)
  2. Chemical peel, microdermabrasion, dermaplaning, or microneedling (time frame 3 months)
  3. Retin-A®, Retin-A Micro®, Renova®, Avita®, Tazorac®, Avage® or Differin® or other similar prescription drugs (time frame 3 months)
  4. Cosmetic injections (filler and/or toxins, i.e. Juvederm, Radiesse, Botox, etc.), non-ablative laser or fractional laser resurfacing (time frame 12 months)
  5. Accutane® or other oral retinoid, Ablative procedures (i.e. laser, chemical) (time frame 12 months)
* Individuals who have any planned surgeries or procedures during the study.
* Individuals who participated in a facial usage study within the last 30 days, or who are currently participating on another usage study.
* Individuals currently on or planning to participate on any type of research study at another facility or a doctor's office during this study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female Caucasian subjects with Fitzpatrick skin types I-III that meet one of the criteria listed; ages 18-30 years old without acne scars on the face with or without visible cellulite on posterior thigh, or ages 55-75 years old without acne scars on the face with or without visible cellulite on posterior thigh, or ages 18-75 years old with atrophic acne scars.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2018-12-07 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
VivoSight software measurements of Epidermal Thickness | Day 1
  Epidermal thickness will be measured in microns.
VivoSight software measurements of surface roughness | Day 1
  Surface roughness measurements (Ra, Rq, Rz) will be measured in microns.
VivoSight software measurements of redness | Day 1
  Redness will be measured in percent
VivoSight software measurements of attenuation coefficient | Day 1
  Attenuation coefficient will be measured in AU (arbitrary unit)

SECONDARY OUTCOMES:
Overall Photodamage Score at Day 1 | Day 1
  The Investigator will assess the participant's overall photodamage using a 10-point scale where (0) = None to (9) = Severe).
Overall Appearance of Fine Lines/Wrinkles Cheek Areas | Day 1
  The investigator will assess the participant's appearance of fine lines/wrinkles using a 5-point scale from (0=None to 4=Diffuse).
Post-study Dynamic Optical Coherence Tomography (D-OCT) Image Analysis of Epidermal Thickness | Day 1
  Post-study D-OCT image analysis will be done (at the sponsor's discretion) by an independent physician expert.
Post-study D-OCT Image Analysis of Density and Attenuation Coefficient of Epidermis | Day 1
  Post-study D-OCT image analysis will be done (at the sponsor's discretion) by an independent physician expert.
Post-study D-OCT Image Analysis of Density and Attenuation Coefficient of Superficial Dermis | Day 1
  Post-study D-OCT image analysis will be done (at the sponsor's discretion) by an independent physician expert.
Post-study D-OCT Image Analysis of Collagen Fibers | Day 1
  Post-study D-OCT image analysis will be done (at the sponsor's discretion) by an independent physician expert. Measured as normal or in bundles.
Post-study D-OCT Image Analysis of Integrity of Collagen | Day 1
  Post-study D-OCT image analysis will be done (at the sponsor's discretion) by an independent physician expert. Measure as (few, moderate, or many fragments).
Post-study D-OCT Image Analysis of Score of Vessels | Day 1
  Post-study D-OCT image analysis will be done (at the sponsor's discretion) by an independent physician expert. Measured at 300 and 500 microns.
Post-study D-OCT Image Analysis of Vascularity Quantification with Thresholds | Day 1
  Post-study D-OCT image analysis will be done (at the sponsor's discretion) by an independent physician expert. Measured at 300 and 500 microns depth.
Blinded Independent Physician Assessor Grading of the D-OCT Images of Stratum Corneum Reflectivity | Day 1
  Grading (0 = absent to 3 = high).
Blinded Independent Physician Assessor Grading of the D-OCT images of Upper Dermal Reflectivity | Day 1
  Grading (0 = absent to 3 = high).
Blinded Independent Physician Assessor Grading of the D-OCT Images of Dermoepidermal Contrast | Day 1
  Grading (0 = absent to 3 = high).
Blinded Independent Physician Assessor Grading of the D-OCT images of Vessel Density | Day 1
  Grading (0 = no vessels to 3 = many vessels).
Antera 3D Images | Day 1
  The investigator will capture 3D images utilizing the Antera 3D.
VISIA-CR Images | Day 1
  The investigator will capture standardized digital photographs utilizing the VISIA-CR.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Goberdhan, Principal Investigator — Allergan
Locations (1):
- Skinmedica Clinical Research and Innovation Center, Irvine, California, United States